CLINICAL TRIAL: NCT07187986
Title: Effectiveness of Sound Acupuncture in Painful Chemotherapy-Related Neuropathies: A Non-Invasive Alternative to Acupuncture? Pilot Study
Brief Title: Sound Acupuncture in Painful Chemotherapy-Related Neuropathies
Acronym: SUONO-PT 01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ente Ospedaliero Ospedali Galliera (Other)
Responsible Party: Principal Investigator, Andrea Assini, MD, Ente Ospedaliero Ospedali Galliera
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 67UCS2018
Record Dates: First submitted 2025-08-04; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Neuropathic Pain in Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sound acupuncture (Experimental): Best medical therapy + Sound Acupuncture
  Interventions: Other: Sound acupuncture
- BMT (No Intervention): Best medical therapy

INTERVENTIONS:
Other: Sound acupuncture — Best medical therapy + soundpuncture
  Arms: Sound acupuncture

SUMMARY:
The objective of this clinical trial is to evaluate the efficacy of sound acupuncture in combination with traditional medical therapy in the treatment of chemotherapy-induced peripheral neuropathies.

Sound acupuncture is a non-invasive technique that involves stimulating energy points, used in acupuncture, with the help of specific tuning forks and the frequencies they emit.

The energy points are those used in Chinese medicine and, more specifically, in acupuncture.

The aim is to restore the recipient's complex bioenergetic system to an optimal state of well-being and balance

Participants:

20 patients will receive only the best medical therapy; 20 patients will receive BMT and sound acupuncture treatment

ELIGIBILITY:
Inclusion Criteria:

* Age 30-80 years
* Clinical and electrophysiological diagnosis of chemotherapy-induced neuropathy
* Patients being treated with Best Medical Therapy for neuropathic pain
* Written informed consent

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Patients with intellectual disabilities or cognitive impairment that impair their ability to comply with the consent process
* Pacemaker users

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-16 (Actual)

PRIMARY OUTCOMES:
Pain reduction | 1 year
  At least a 30% reduction from baseline on the NPS scale for neuropathic pain

SECONDARY OUTCOMES:
Back Depression inventory | 1 year
  Effectiveness of sound therapy combined with pharmacological treatment through administration of the BDI-II scale
Quality of life assessment | 1 year
  EQ-5D scale for assessing the impact on quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- E.O. Ospedali Galliera, Genoa, Liguria, Italy